CLINICAL TRIAL: NCT01019044
Title: Virologic and Immunologic Evaluation of the Deep Viral Reservoirs in HIV-1 Infected Patients With Long Term Viral Suppression
Brief Title: Exploration of HIV Reservoirs
Acronym: MUCOVIR
Status: Completed | Type: Observational
Sponsor: Objectif Recherche Vaccins SIDA (Other)
Responsible Party: Sponsor
Other Study IDs: ORVACS 009
Record Dates: First submitted 2009-11-24; First posted 2009-11-25 (Estimated); Last update posted 2013-02-13 (Estimated); Status verified 2013-02

CONDITIONS: HIV-1 Infection
Keywords: HIV; Viral reservoirs; Viral load

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — Plasma and total blood samples A maximum of 15 rectal mucosa biopsy samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Rectal mucosa biopsy: Rectal mucosa samples collection
  Interventions: Procedure: Rectal mucosa biopsy

INTERVENTIONS:
Procedure: Rectal mucosa biopsy — Collection of a maximum of 15 rectal mucosa samples in the high portion of the rectum near the rectosigmoidal junction

SUMMARY:
Prospective study in HIV-1 infected patients with a plasma viral load below the limit of detection and stable for at least 5 years.

DETAILED DESCRIPTION:
Evaluation of the mucosal HIV reservoirs (HIV-DNA quantification and distribution of the infected T lymphocytes in the gut mucosa associated lymphoid tissue compared to the blood in HIV-1 infected patients under antiretroviral treatment with an undetectable plasma viral load below the 50 copies/ml limit of detection for at least 5 years).

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 documented infection
* HIV-1 plasma viral load measurable before antiretroviral treatment initiation
* Patients treated with an antiretroviral combination containing a protease inhibitor and/or a non-nucleosidic reverse transcriptase inhibitor without any interruption since treatment initiation
* Patients with a stable plasma viral load below the limit of detection (HIV-RNA < 50 copies/ml since January 2006 and/or HIV-RNA < 200 copies/ml during the anterior period) under antiretroviral treatment for at least 5 years and for at least 90 % of the measures

Exclusion Criteria:

* Contraindication to the biopsy
* No ability or willingness to provide informed consent
* Concomitant treatment with antithrombotics or platelets antiaggregatory
* Patients co-infected with HCV and or HBV
* Patients who received an immunosuppressive treatment during 3 months prior enrollment (chemotherapy, radiotherapy, corticotherapy, splenectomy) or an immunotherapy during 5 years prior enrolment (IL-2, anti-HIV vaccine, IFN-alpha)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV-1 infected patients followed in specialized infectious disease/HIV hospital department
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2009-05; Primary Completion 2009-10 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Quantification of the HIV-RNA plasma viral load using ultrasensible assay (limit of detection: 1 copy/ml) | Single patient visit

SECONDARY OUTCOMES:
Quantification of the HIV proviral DNA in the rectal mucosa biopsies and in the PPBMCs | Single patient visit
Quantitative, phenotypic and functional description of the long-term immune reconstitution in the rectal mucosa biopsies | Single patient visit
Quantification of HIV proviral DNA in the total CD4 lymphocytes | Single patient visit
Pharmacokinetics of the antiretroviral molecules in the rectal mucosa biopsies and in the blood | Single patient visit

CONTACTS AND LOCATIONS:
Overall Officials: Christine KATLAMA, MD, Principal Investigator — Groupe Hospitalier Pitié-Salpêtrière; François LECARDONNEL, MSc, Study Director — ORVACS
Locations (1):
- Groupe Hospitalier Pitié-Salpêtrière, Paris, France

REFERENCES:
- [Result] Descours B, Lambert-Niclot S, Mory B, Samri A, Charlotte F, Peytavin G, Tubiana R, Papagno L, Bacchus C, Lecardonnel F, Katlama C, Autran B, Marcelin AG, Valantin MA, Carcelain G; DECAMUNE and ORVACS Study Groups. Direct quantification of cell-associated HIV DNA in isolated rectal and blood memory CD4 T cells revealed their similar and low infection levels in long-term treated HIV-infected patients. J Acquir Immune Defic Syndr. 2013 Mar 1;62(3):255-9. doi: 10.1097/QAI.0b013e318282537f. PMID 23274932